CLINICAL TRIAL: NCT05875272
Title: Prospective, Monocentric Study of the Interchangeability of Arterial Coagulation and Venous Coagulation, in the Context of Cardiac Surgeries Under Cardiopulmonary Bypass, Using the DMDiv Hemochron Signature Elite
Brief Title: Interchangeability of Arterial Coagulation and Venous Coagulation, in the Context of Cardiac Surgeries Under Cardiopulmonary Bypass, Using the DMDiv Hemochron Signature Elite
Acronym: COAGAV
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0057
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hemostasis; Extracorporeal Circulation; Heparin; Cardio-pulmonary Bypass
Keywords: Hemostasis; extra corporeal circulation; heparin; Activated Clotting Time; Hemochron; venous and arterial blood; cardio-pulmonary bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: interchangeability of arterial or venous hemostasis — Paired arterial and venous blood sampling respectively on the radial arterial catheter and on the central venous catheter before the extracorporeal circulation, and on the sampling ramp during the extracorporeal circulation. Point of care biology exams are performed on two HSE devices simultaneously. Controls carried out, routinely, every 20 minutes according to the service protocol, before the CPB (starting ACT without heparin), during the CPB (ACT objective ≥400 seconds), after protamine reversal of heparin. On average, 10 samples are taken during heart surgery.

SUMMARY:
Adequate coagulation measured using activated clotting (ACT) is important during vascular and cardiac surgeries. Unfractionated heparin is the most common anticoagulant used. For point of care testing, under supervision of biology department, the investigators use Hemochron Signature Elite®(HSE) (Werfen®-Barcelona Spain) to determine coagulation during cardiac surgery under Cardiopulmonary Bypass (CPB), with arterial or venous blood. The dosage of heparin varies according to this result, throughout the CPB. On the Connect Manager® software (Livanova®, Italy) which records all the data of a CPB, it is mandatory to inform, during an ACT, the sampling site in arterial or venous. The chemical compositions of arterial blood and venous blood are different (O2, Co2…) Even if the qualities of coagulation in vivo are identical, what happens when they are chemically analyzed using the medical device HSE ? Can we trust the results of this device to secure anticoagulation under CPB? Are the results affected by the sampling site? The objective of this study is to compare the reliability of hemostasis control , during cardiac surgery under cardiopulmonary bypass, for both venous and arterial blood. Effective and controllable anticoagulation is mandatory during cardiac surgeries under extracorporeal circulation. The monitoring of the effectiveness of heparin is carried out, in our center, using the Hemochron Signature Elite® (HSE) medical device, which measures the ACT (Activated Clotting Time). There is no comparative study between hemostasis of venous blood, versus arterial blood, with this point of care device.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over,
* undergoing conventional heart surgery under normothermic Cardiopulmonary Bypass (nadir 34°) (Aortic valve replacement, coronary artery bypass graft surgery, valve plasty, atrial septal defect, ventricular septal defect, intracardiac tumours, heart surgery, ascending aorta, combined surgery…)
* They must be affiliated with Social Security in France, and have given their written consent.

Exclusion Criteria:

* Minor Patients,
* Emergency Cardiac Surgeries, Extracorporeal circulation in hypothermia, Cardiac surgery without CEC
* Patients already included in a research protocol,
* Patient under guardianship or curators or deprived of public law,
* Patient with proven Heparin Induced Thrombopenia (HIT) not receiving heparin
* Pregnant woman, breastfeeding or parturient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and over, undergoing conventional heart surgery under normothermic Cardiopulmonary Bypass (nadir 34°) (Aortic valve replacement, coronary artery bypass graft surgery, valve plasty, atrial septal defect, ventricular septal defect, intracardiac tumours, heart surgery, ascending aorta, combined surgery…)
Sampling Method: Non-Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Activated Clotting Time after using the Hemochron Signature Elite® medical device | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No